CLINICAL TRIAL: NCT02342106
Title: Assessment of Myeloid Cell Constitution in the Follicular Fluid of Women Undergoing In-vitro Fertilization (IVF)
Brief Title: Assessment of Myeloid Cell Constitution in the Follicular Fluid of Women Undergoing In-vitro Fertilization
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0054-14-HYMC
Record Dates: First submitted 2014-12-28; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Follicular fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Poor responders: In order to define the poor response in IVF, at least two of the following three features must be present: (i) advanced maternal age or any other risk factor for poor ovarian response; (ii) a previous poor ovarian response; and (iii) an abnormal ovarian reserve test . Two episodes of poor ovarian response after maximal stimulation are sufficient to define a patient as poor responder in the absence of advanced maternal age or abnormal ovarian reserve test. By definition, the term poor ovarian response refers to the ovarian response, and therefore, one stimulated cycle is considered essential for the diagnosis .
- Good responders: Total number of antral follicles : 22-35 Normal (good) antral count, should have an excellent response to ovarian stimulation.Likely to respond well to low doses of FSH drugs.
  Very low risk for IVF cycle cancellation. Some risk for ovarian overstimulation if a Lupron trigger is not used for final egg maturation injection.
  Excellent pregnancy success rates.

SUMMARY:
The investigators will study the immune cell subpopulations in follicular fluid of patients undergoing In-Vitro Fertilization (IVF) treatment in our clinic. The investigators will corelate the presence of immature myeloid cells to the ovarian stimulation response as indicated by follicle stimulating hormone (FSH) and number of follicles or estradiol level developed on the day of human chorionic gonadotropin (hCG) administration.

DETAILED DESCRIPTION:
The study will be an observational study using discarded material from patients undergoing IVF treatment. On the day of ovum pick up, the fluid aspirated from the first follicle in each ovary will be saved and analyzed for cellular content by fluorescence-activated cell sorter (FACS) analysis and cytokine and hormone by Enzyme-linked immunosorbent assay (ELISA) and quantitative polymerase chain reaction (qPCR). In addition, a total of 5cc of blood will be drawn from the patient when introducing the intravenous line for analysis of immune cell composition,hormones and cytokine levels. During the whole study number of oocytes retrieved,number of mature oocytes,number of fertilizations,implantation rates and clinical pregnancy rates will be documented as well.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF treatment
* Infertility caused by one of the following : endometriosis, severe male factor, tubal occlusion, or unexplained.

Exclusion Criteria:

* An early follicular phase (day 2-4) FSH level > 20 mIU/mL
* Abnormal uterine cavity
* Any contraindication for pregnancy
* Systemic disease
* History of alcohol or drug abuse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing IVF treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-08 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Amount of immature myeloid cells accumulate in the ovarian follicular fluid as measure of correlation with ovarian response to gonadotropins. | 36 hours after hCG injection
  After oocyte retrieval, the fluid of the largest follicle in each ovary will be collected. Follicular fluid cells will be isolated and immunostained for flow cytometry using monoclonal antibodies and the amount of immature myeloid cell will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Limonad, MD, Principal Investigator — Hillel Yaffe Medical Center Hadera Israel
Locations (1):
- Department of Obstetrics and Gynecology, Hillel-Yaffe Medical Center, Hadera, Israel